CLINICAL TRIAL: NCT02469389
Title: Improving Negative Symptoms & Community Engagement in Veterans With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1293-R; NCT02455349 (obsolete NCT alias)
Record Dates: First submitted 2015-06-08; First posted 2015-06-11 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Schizophrenia; Serious Mental Illness
Keywords: Schizophrenia; Negative Symptoms
MeSH Terms: conditions — Schizophrenia | interventions — enc protein, Drosophila; Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Engaging in Community Roles and Experiences (ENCoRE) (Experimental): Engaging in Community Roles and Experiences (ENCoRE) includes evidence-based psychosocial treatment strategies to target the affective-motivational deficits, negative expectancies, and behavioral skills deficits that are central to the maintenance of negative symptoms. Behavioral strategies include motivational enhancement, psychoeducation, cognitive therapy, and social skills training.
  Interventions: Behavioral: Engaging in Community Roles and Experiences (ENCoRE)
- Health & Wellness (H&W) (Active Comparator): Health & Wellness (H&W) will focus on health and wellness issues and education on ways to better manage health-related concerns following a basic structure that includes: review of the previous session's material, new educational content, and discussion/application. Topics will include: 1) Overview, 2) Physical Activity (3 sessions), 3) Nutrition/Healthy Eating (3 sessions), 4) Managing Fatigue/Sleep (3 sessions), 5) Relaxation (3 sessions), 6) Tobacco cessation (3 sessions), 7) Substance Use (3 sessions), 8) Medication/Side Effects (3 sessions), 9) Review (1 session), and Closing (1session).
  Interventions: Behavioral: Health & Wellness (H&W)

INTERVENTIONS:
Behavioral: Engaging in Community Roles and Experiences (ENCoRE) — Engaging in Community Roles and Experiences (ENCoRE) includes evidence-based psychosocial treatment strategies to target the affective-motivational deficits, negative expectancies, and behavioral skills deficits that are central to the maintenance of negative symptoms. Behavioral strategies include motivational enhancement, psychoeducation, cognitive therapy, and social skills training.
  Other Names: ENCoRE
  Arms: Engaging in Community Roles and Experiences (ENCoRE)
Behavioral: Health & Wellness (H&W) — Health & Wellness (H&W) will focus on health and wellness issues and education on ways to better manage health-related concerns following a basic structure that includes: review of the previous session's material, new educational content, and discussion/application.
  Topics will include: 1) Overview, 2) Physical Activity (3 sessions), 3) Nutrition/Healthy Eating (3 sessions), 4) Managing Fatigue/Sleep (3 sessions), 5) Relaxation (3 sessions), 6) Tobacco cessation (3 sessions), 7) Substance Use (3 sessions), 8) Medication/Side Effects (3 sessions), 9) Review (1 session), and Closing (1session).
  Other Names: H&W
  Arms: Health & Wellness (H&W)

SUMMARY:
The goal of this project is to evaluate an innovative psychosocial intervention package that will incorporate evidence-based treatment strategies to target the affective-motivational deficits, negative expectancies, and behavioral skills deficits that are central to the maintenance of negative symptoms. The intervention - called EnCoRE (Engaging in Community Roles and Experiences) - will include strategies aimed at teaching Veterans with schizophrenia and negative symptoms ways to (1) overcome deficits in anticipatory pleasure, (2) increase intrinsic motivation for goal-directed activities, (3) reduce expectancies for failure, and (4) perform skillfully in new social situations, all of which can impact implementation of new skills and behaviors. Rather than develop a new set of intervention strategies, the investigators will include within EnCoRE evidence-based strategies for these treatment domains. In addition, the investigators will collect qualitative information both from Veterans concerning their perceptions of the strengths, weaknesses, and barriers to participation in EnCoRE, as well as from a sample of mental health providers who work with Veterans with schizophrenia and negative symptoms, in order to inform a larger scale implementation trial should EnCoRE prove effective here.

DETAILED DESCRIPTION:
The goal of this study is to evaluate an innovative psychosocial intervention package that will incorporate evidence-based treatment strategies to target the affective-motivational deficits, negative expectancies, and behavioral skills deficits that are central to the maintenance of negative symptoms. The intervention - called EnCoRE (Engaging in Community Roles and Experiences) - will include strategies aimed at teaching Veterans with schizophrenia and negative symptoms ways to (1) overcome deficits in anticipatory pleasure, (2) increase intrinsic motivation for goal-directed activities, (3) reduce expectancies for failure, and (4) perform skillfully in new social situations, all of which can impact implementation of new skills and behaviors. Rather than develop a new set of intervention strategies, the investigators will include within EnCoRE evidence-based strategies for these treatment domains. In addition, the investigators will collect qualitative information both from Veterans concerning their perceptions of the strengths, weaknesses, and barriers to participation in EnCoRE, as well as from a sample of mental health providers who work with Veterans with schizophrenia and negative symptoms, in order to inform a larger scale implementation trial should EnCoRE prove effective here.

Following a short pilot to train interventionists and refine the manual, the investigators will conduct a randomized controlled trial to test the efficacy of EnCoRE in improving ratings of negative symptoms, functional outcomes, and engagement in community activities in a sample of Veterans with schizophrenia and negative symptoms (n=108). Participants will be randomized either to EnCoRE or a health-related control group. These goals fit well within the objectives of the Rehabilitation Research and Development (RR&D) program of funding research aimed at studying rehabilitation interventions focused on maximizing functional recovery and assisting in the integration of Veterans into civilian life. Specifically, the investigators will address the following Specific Aims:

Specific Aim 1: Train therapists and refine the EnCoRE manual in a preliminary trial with 10 Veterans with schizophrenia and negative symptoms.

Specific Aim 2: Conduct a randomized controlled trial (n=108, medium effect, alpha=.05) to test the efficacy of EnCoRE in producing positive changes at post-treatment and 3-month follow-up on the primary outcomes of negative symptoms and social and community functioning.

Specific Aim 3: Examine qualitative interviews completed by (1) Veterans who participated in EnCoRE and (2) Mental Health Providers to determine aspects of EnCoRE that were perceived as more or less helpful, interesting, and valuable in order to make adjustments prior to conducting a larger, multi-site implementation trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Disorders, 5th edition (DSM 5) diagnosis of schizophrenia or schizoaffective disorder
* A minimum average rating of a "moderately severe deficit" (3 or greater on a 0-4 scale) on one symptom domain or a minimum average rating of a "moderate deficit" (2 or greater on a 0-4 scale) on two or more domains, within the affect motivation factor of the Clinical Assessment Interview for Negative Symptoms (CAINS) i.e.,:

  * symptoms of asociality
  * avolition
  * anhedonia
* Age between 18 and 75 years
* Seen by a service provider twice within the last 6 months or once in the last 6 months consistently for two years, as in line with the Veteran's recorded mental health treatment plan (to demonstrate that participants receive ongoing and regular mental health care)
* Competent to sign Informed Consent

Exclusion Criteria:

* Documented history of serious neurological disorder or head trauma with loss of consciousness
* Cognitive impairment (defined as a total intelligence quotient (IQ) score less than 70 as measured by the Wechsler Test of Adult Reading or as indicated by chart review
* Inability to effectively participate in the baseline assessments due to psychiatric symptoms on two successive appointments
* Current problematic substance use as indexed by scores on the Michigan Alcoholism Screening Test and the Drug Abuse Screening Test
* Currently meet criteria for a major depressive episode

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie E Bennett, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bennett ME, Kuykendall L, Harvey K, Lucksted A. Increasing community engagement: Skills used by adults with schizophrenia participating in a psychosocial intervention. Psychiatr Rehabil J. 2023 Mar;46(1):83-93. doi: 10.1037/prj0000549. PMID 36809019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial took place at three mid-Atlantic VA Medical Centers; participants were recruited between 12/10/2015 and 7/25/2019.
Pre-assignment Details: 154 individuals signed consent to participate. Of these, 49 were not randomized due to: (1) 41 did not pass eligibility screening; (2) 7 did not complete screening; (3) 1 did not complete the baseline assessment.
Groups:
- Health & Wellness (H&W): Health & Wellness (H&W) will focus on health and wellness issues and education on ways to better manage health-related concerns following a basic structure that includes: review of the previous session's material, new educational content, and discussion/application. Topics will include: 1) Overview, 2) Physical Activity (3 sessions), 3) Nutrition/Healthy Eating (3 sessions), 4) Managing Fatigue/Sleep (3 sessions), 5) Relaxation (3 sessions), 6) Tobacco cessation (3 sessions), 7) Substance Use (3 sessions), 8) Medication/Side Effects (3 sessions), 9) Review (1 session), and Closing (1session).
  Health & Wellness (H&W): Health & Wellness (H&W) will focus on health and wellness issues and education on ways to better manage health-related concerns following a basic structure that includes: review of the previous session's material, new educational content, and discussion/application.
  Topics will include: 1) Overview, 2) Physical Activity (3 sessions), 3) Nutrition/Healthy Eating (3 sessions), 4) Managing Fatigue/Sleep (3 sessions), 5) Relaxation (3 sessions), 6) Tobacco cessation (3 sessions), 7) Substance Use (3 sessions), 8) Medication/Side Effects (3 sessions), 9) Review (1 session), and Closing (1session).
Period: Overall Study
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Started | 53 | 52
Completed 12-week Assessment | 40 (13 lost to contact or refused) | 44 (8 lost to contact or refused)
Completed 24-week Assessment | 37 (16 lost to contact or refused) | 46 (6 lost to contact or refused)
Completed | 37 | 44
Not Completed | 16 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W) | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (11.7) | 57.6 (9.1) | 55.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 47 | 49 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 53 | 50 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 36 | 78
  White | 8 | 10 | 18
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Diagnosis [Count of Participants; unit: Participants] — Type of schizophrenia spectrum disorder as assessed via a structured diagnostic interview
  Participants
    Schizophrenia | 20 | 30 | 50
    Schizoaffective disorder | 33 | 22 | 55

OUTCOME MEASURES:

1. Primary Outcome: Clinical Assessment Interview for Negative Symptoms Motivation & Pleasure Scale (CAINS MAP) - 12 Weeks
Description: Differences in mean change on the CAINS MAP scale from baseline assessment to 12 week assessment. This scale contains a total of 9 items, each with a range of 0-4. Scores range from 0-36. Lower scores mean a better outcome.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 12 weeks
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  Baseline | 19.8 (5.1) | 17.3 (4.8)
  12 week assessment | 17.4 (5.8) | 17.1 (4.9)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Analyses of the primary and secondary outcomes utilized a linear mixed effects model accounting for random therapy group effects and included all available data at baseline (BL), post-treatment (PT; 12-week), and follow-up (FU; 24-week) timepoints (TPs). Error terms across TPs were assumed correlated with unstructured correlation matrix. To test time specific hypotheses, terms in the mean model included separate indicators for PT & FU & interaction terms between these indicators and conditions; Test type: Superiority — Based on randomization to treatment condition, the model assumed no differences at BL (any difference was assumed due to random sampling error); p = 0.295, Mixed Models Analysis; Post-hoc mixed effects model analyses of all outcomes were performed adjusting for BL CAINS MAP score

2. Primary Outcome: Social Functioning Scale (SFS) - 12 Weeks
Description: Differences in mean change on the SFS from baseline assessment to 12 week assessment. In the present analysis, we used a total score for the SFS including all subscales except the employment subscale. Scores ranged from 13-213. Higher scores mean a better outcome.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 12 weeks
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  SFS at baseline assessment | 110.3 (20.8) | 114.0 (19.5)
  SFS at 12 week assessment | 111.1 (19.5) | 112.1 (112.1)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Test type: Superiority; p = 0.182, Mixed Models Analysis

3. Primary Outcome: Clinical Assessment Interview for Negative Symptoms Motivation & Pleasure Scale (CAINS MAP) - 24 Weeks
Description: Differences in mean change on the CAINS MAP scale from baseline assessment to 24 week assessment. This scale contains a total of 9 items, each with a range of 0-4. Scores range from 0-36. Lower scores mean a better outcome.
Time Frame: Participants will be assessed a second time following completion of the study intervention, an expected average of 24 weeks
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  CAINS MAP at baseline assessment | 19.8 (5.1) | 17.3 (4.8)
  CAINS MAP at 24 week assessment | 16.2 (6.1) | 17.2 (5.3)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Test type: Superiority; p = 0.114, Mixed Models Analysis

4. Primary Outcome: Social Functioning Scale (SFS) - 24 Weeks
Description: Differences in mean change on the SFS from baseline assessment to 24 week assessment. In the present analysis, we used a total score for the SFS including all subscales except the employment subscale. Scores ranged from 13-213. Higher scores mean a better outcome.
Time Frame: as for outcome 3
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  SFS at baseline | 110.3 (20.8) | 114.0 (19.5)
  SFS at 24 week assessment | 116.8 (26.5) | 112.7 (20.4)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Test type: Superiority; p = 0.220, Mixed Models Analysis

5. Secondary Outcome: University of California San Diego Performance Based Skills Assessment - Brief (UPSA-B) - 12 Weeks
Description: Differences in mean change on the UPSA-B from baseline assessment to 12 week assessment. The UPSA-B has a range of 0-100 with higher scores mean a better outcome. In the present analysis, we used the square root of UPSA-B scores with range 0-10.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 12 weeks
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  UPSA-B at baseline | 8.5 (1.0) | 8.4 (1.2)
  UPSA-B at 12 week assessment | 8.7 (0.8) | 8.1 (1.3)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Test type: Superiority; p = 0.018, Mixed Models Analysis

6. Secondary Outcome: Maryland Assessment of Recovery Scale (MARS) - 12 Weeks
Description: Differences in mean change on the MARS from baseline assessment to 12 week assessment. Scores can range from 25-125. Higher scores mean a better outcome.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 12 weeks
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  MARS score at baseline | 95.5 (16.0) | 96.7 (17.7)
  MARS score at 12 week assessment | 95.0 (18.2) | 96.1 (19.4)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Test type: Superiority; p = 0.903, Mixed Models Analysis

7. Secondary Outcome: Clinical Assessment Interview for Negative Symptoms Social Motivation and Pleasure Subscale (CAINS SMAP) - 12 Weeks
Description: Differences in mean change on the CAINS SMAP from baseline assessment to 12 week assessment. This subscale has a total of 4 items each rated on a 0-4 score. The range of scores was 0-16. Lower scores mean a better outcome.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 12 weeks
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  SMAP rating at baseline | 8.6 (3.4) | 7.1 (3.7)
  SMAP rating at 12 week assessment | 6.9 (3.7) | 6.8 (3.4)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Test type: Superiority; p = 0.535, Mixed Models Analysis

8. Secondary Outcome: Role Functioning Scale (RFS) - 12 Weeks
Description: Differences in mean change on the RFS from baseline assessment to 12 week assessment. Items are rated on a 1 to 7 scale. In the present analysis, we summed ratings of Family Network Relationships and Immediate Social Network Relationships as our measure of role functioning. Scores can range from 2-14. Higher scores mean a better outcome.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 12 weeks
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  RFS at baseline | 9.0 (2.8) | 8.9 (3.1)
  RFS at 12 week assessment | 11.0 (2.7) | 9.5 (2.6)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Test type: Superiority; p = 0.010, Mixed Models Analysis

9. Secondary Outcome: University of California San Diego Performance Based Skills Assessment - Brief (UPSA-B) - 24 Weeks
Description: Differences in mean change on the UPSA-B from baseline assessment to 24 week assessment. The UPSA-B has a range of 0-100 with higher scores mean a better outcome. In the present analysis, we used the square root of UPSA-B scores with range 0-10.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 24 weeks
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  UPSA-B score at baseline | 8.5 (1.0) | 8.4 (1.2)
  UPSA-B score at 24 week assessment | 8.6 (0.8) | 8.6 (0.9)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Test type: Superiority; p = 0.692, Mixed Models Analysis

10. Secondary Outcome: Maryland Assessment of Recovery Scale (MARS) - 24 Weeks
Description: Differences in mean change on the MARS from baseline assessment to 24 week assessment. Scores can range from 25-125. Higher scores mean a better outcome.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 24 weeks
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  MARS score at baseline | 95.5 (16.0) | 96.7 (17.7)
  MARS score at 24 week assessment | 95.8 (17.9) | 95.5 (19.2)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Test type: Superiority; p = 0.498, Mixed Models Analysis

11. Secondary Outcome: Clinical Assessment Interview for Negative Symptoms Social Motivation and Pleasure Subscale (CAINS SMAP) - 24 Weeks
Description: Differences in mean change on the CAINS SMAP from baseline assessment to 24 week assessment. This subscale has a total of 4 items each rated on a 0-4 score. The range of scores was 0-16. Lower scores mean a better outcome.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 24 weeks
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  CAINS SMAP score at baseline | 8.6 (3.4) | 7.1 (3.7)
  CAINS SMAP score at 24 week assessment | 6.4 (3.7) | 7.6 (3.6)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Test type: Superiority; p = 0.079, Mixed Models Analysis

12. Secondary Outcome: Role Functioning Scale (RFS) - 24 Weeks
Description: Differences in mean change on the RFS from baseline assessment to 24 week assessment. Items are rated on a 1 to 7 scale. In the present analysis, we summed ratings of Family Network Relationships and Immediate Social Network Relationships as our measure of role functioning. Scores can range from 2-14. Higher scores mean a better outcome.
Time Frame: Participants will be assessed following completion of the study intervention, an expected average of 24 weeks
Population: All participants randomized to study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
Number analyzed (Participants) | 53 | 52
score on a scale
  RFS at baseline | 9.0 (2.8) | 8.9 (3.1)
  RFS at 24 week assessment | 10.4 (2.7) | 9.7 (2.8)
Statistical Analysis 1: Comparison: Engaging in Community Roles and Experiences (ENCoRE) vs Health & Wellness (H&W); Test type: Superiority; p = 0.539, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 5 years
Description: All Serious Adverse Events were medical or psychiatric hospitalizations. All Other Adverse Events were emergency room visits for medical or psychiatric problems that did not result in hospitalization.
Arm/Group | Engaging in Community Roles and Experiences (ENCoRE) | Health & Wellness (H&W)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 9/53 | 7/52
Other Adverse Events (participants affected / at risk) | 4/53 | 5/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engaging in Community Roles and Experiences (ENCoRE) (N=53) | Health & Wellness (H&W) (N=52)
Hospitalization (General disorders) | 9 (11) | 7 (8) — Hospitalization for a medical or psychiatric disorder
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engaging in Community Roles and Experiences (ENCoRE) (N=53) | Health & Wellness (H&W) (N=52)
Emergency room visits (General disorders) | 4 (4) | 5 (6) — Emergency room visits for medical or psychiatric disorders

LIMITATIONS AND CAVEATS:
Target sample size=108 (we randomized 105) to achieve 80% power to detect a Cohen's d type effect size at 12 weeks=0.50 ("medium") on primary outcomes. This may have been too large an effect to expect for a behavioral intervention with an active control; the study may have been underpowered. The arms differed on BL CAINS MAP. We reran all mixed model analyses adjusting for BL CAINS MAP. Results remained the same except the difference in mean change on the CAINS SMAP at FU was significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT02469389/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT02469389/SAP_001.pdf